# STATISTICAL ANALYSIS PLAN (SAP)

# **SM04690-OA-06 – Phase B**

**Study Title:** A Phase 2, 52-Week, Multicenter, Randomized, Double-Blind,

Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of Two Injections of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis

Subjects

**Protocol Number:** SM04690-OA-06

**Protocol Version:** Amendment 04 Version 00, 21 August 2020

**SAP Version:** 00, 22 September 2021

**Investigational Product:** SM04690 Injectable Suspension

Clinical Phase: Phase 2

This document is the sole property of Biosplice Therapeutics, Inc. This document and any and all information contained herein must be considered and treated as strictly confidential. This document shall be used only for the purpose of the disclosure herein provided. No disclosure or publication shall be made without the prior written consent of Biosplice Therapeutics, Inc.

Phase B SAP Version 00 22 September 2021

# SIGNATURE PAGE AND APPROVALS

A Phase 2, 52-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of Two Injections of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects

**Protocol Version:** Amendment 04 Version 00, 21 August 2020

**SAP Version:** Version 00

Date: 22 September 2021

| Name & Title | Signature | Date |
|---|---|---|
| Jonathan Britt, M.S. | Document has been electronically sign | |
| Manager, Biostatistics | final page of the viewable rendition for electronic signature(s). | |
| Christopher Swearingen, Ph.D. | Document has been electronically sign final page of the viewable rendition for | |
| Vice President, Biometrics | signature(s). | relectronic |
| Ismail Simsek, M.D. | Document has been electronically sign final page of the viewable rendition for | |
| Medical Director | signature(s). | electronic |
| Amy Halseth, Ph.D. | Document has been electronically sign | ned. Please see the |
| Executive Director, Clinical Science | final page of the viewable rendition for electronic signature(s). | |

Biosplice Therapeutics commits to satisfying the requirements of the International Council for Harmonisation Good Clinical Practice (ICH-GCP) Guidelines regarding the responsibilities of the Sponsor, the United States (US) Code of Federal Regulations (CFR) Title 21 Parts 50, 54, 56, 312, and 314, and GCP Guidelines, as applicable.

# TABLE OF CONTENTS

| | | | E PAGE AND APPROVALS | |
|---|-----|-------|----------------------------------------------------|-----|
| T | ABL | LE OF | CONTENTS | 3 |
| A | BBF | REVIA | TIONS | 6 |
| 1 | В | ACKO | GROUND | 8 |
| 2 | 0 | VERV | /IEW | 9 |
| 3 | S | TUDY | OBJECTIVES AND ENDPOINTS | 9 |
| | 3.1 | Stud | ly Objective | 9 |
| | 3. | .1.1 | Primary Objective | 9 |
| | 3. | .1.2 | Secondary Objectives | 9 |
| | 3.2 | Stud | dy Endpoints | . 0 |
| | 3. | .2.1 | Phase A General Safety Endpoints | C |
| | 3. | .2.2 | Phase A Bone Imaging Endpoints | C |
| | 3. | .2.3 | Phase A Efficacy Endpoints | C |
| | 3. | .2.4 | Phase A Exploratory Biomarker Endpoints | . 1 |
| | 3. | .2.5 | Phase B General Safety Endpoints | . 1 |
| | 3. | .2.6 | Phase B Bone Imaging Endpoints | . 1 |
| | 3. | .2.7 | Phase B Efficacy Endpoints | . 1 |
| | 3. | .2.8 | Phase B Exploratory Biomarker Endpoints | . 2 |
| 4 | 0 | VERA | ALL STUDY DESIGN AND PLAN1 | 2 |
| | 4.1 | Sele | ection of Study Population | . 2 |
| | 4.2 | Met | hod of Treatment Assignment and Randomization | . 2 |
| | 4.3 | Trea | atment Blinding | . 2 |
| | 4.4 | Mir | imization of Missing Data | .3 |
| | 4. | .4.1 | Collection of Clinical Outcomes | .3 |
| | 4. | .4.2 | Prohibited Medications, Treatments, and Procedures | .3 |
| | 4. | .4.3 | Intermittent Missing Data | .3 |
| 5 | A | NALY | SIS AND REPORTING1 | 3 |
| | 5.1 | Pha | se A Analysis1 | .3 |
| | 5.2 | Pha | se B Analysis | .3 |
| 6 | S | AMPL | E SIZE DETERMINATION 1 | 3 |

| 7 | AN | ALYSIS POPULATIONS | 14 |
|---|------|-------------------------------------------------------|----|
| | 7.1 | Full Analysis Set | 14 |
| | 7.2 | Full Analysis Set Phase B | 14 |
| | 7.3 | Modified Full Analysis Set | 14 |
| | 7.4 | Per-Protocol Analysis Set | 14 |
| | 7.5 | Per-Protocol Analysis Set Phase B | 14 |
| | 7.6 | Safety Analysis Set | 14 |
| | 7.7 | Safety Analysis Set Phase B. | 14 |
| 8 | GE | NERAL ISSUES FOR STATISTICAL ANALYSIS | 15 |
| | 8.1 | General Statistical Methodology | 15 |
| | 8.1. | 1 Baseline | 15 |
| | 8.1. | .2 Analysis of Covariance (ANCOVA) Section 8.1.2 | 15 |
| | 8.1. | .3 Mixed-Effects Models for Repeated Measures | 15 |
| | 8.1. | .4 Data Handling for Subjects Who Withdrew from Study | 16 |
| | 8.1. | .5 Imputation of Missing Data | 16 |
| | 8.2 | General Safety Assessments | 16 |
| | 8.2. | .1 Adverse Events | 16 |
| | 8.2. | .2 Vital Signs and Weight | 16 |
| | 8.2. | .3 Clinical Laboratory Evaluations | 16 |
| | 8.3 | Bone Imaging Assessments | 17 |
| | 8.3. | .1 Knee BMD (qCT) | 17 |
| | 8.3. | .2 Spine and Hip BMD (DXA) | 17 |
| | 8.4 | Efficacy Assessments | 18 |
| | 8.4. | 1 Pain NRS | 18 |
| | 8.4. | 2 WOMAC | 18 |
| | 8.4. | .3 Patient Global Assessment of Disease Activity | 18 |
| | 8.4. | .4 mJSW | 19 |
| | 8.5 | Exploratory Biomarker Assessments | 19 |
| 9 | STU | UDY SUBJECTS AND DEMOGRAPHICS | 19 |
| | 9.1 | Disposition of Subjects and Withdrawals | 19 |
| | 9.2 | Protocol Deviations Section 9.2 | |
| | 9.3 | Demographics and Other Baseline Characteristics | 20 |

| 9.4 | 1 | Medical History | 21 |
|---|---|---|---|
| 10 | ( | GENERAL SAFETY ANALYSIS | 21 |
| 10. | .1 | Adverse Events | 21 |
| 10. | .2 | Vital Signs and Weight | 21 |
| 10. | .3 | Clinical Laboratory Evaluations | 21 |
| 11 | F | BONE IMAGING ANALYSIS | 22 |
| 12 | F | EFFICACY ANALYSIS Section 12 | 22 |
| 13 | F | EXPLORATORY BIOMARKER ANALYSIS | 23 |
| 14 | N | MEDICATIONS | 23 |
| 14. | .1 | Concomitant Medications | 23 |
| 14. | .2 | Exposure | 23 |
| 15 | ( | CHANGES TO PLANNED ANALYSIS | 24 |
| 16 | F | REFERENCES | 24 |
| 17 | A | APPENDICES | 26 |
| 17. | .1 | Appendix 1 – Visit Windows | 26 |
| 17. | .2 | Appendix 2 – Protocol Deviations Leading to Exclusion from Per-Protocol Analysis. | 29 |

# **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|----------------------------------------------------|
| AE | adverse event |
| ANCOVA | analysis of covariance |
| β-СТХ | β-C-terminal telopeptide |
| BMD | bone mineral density |
| CV | coefficient of variation |
| COMP | cartilage oligomeric matrix protein |
| DXA | dual-energy x-ray absorptiometry |
| eCRF | electronic case report form |
| EOSa | Phase A End of Study |
| EOSb | Phase B End of Study |
| ET | early termination |
| FAS | Full Analysis Set |
| FASB | Full Analysis Set Phase B |
| MAR | missing at random |
| mFAS | Modified Full Analysis Set |
| MMRM | mixed-effects model for repeated measures |
| mJSW | medial joint space width |
| OA | osteoarthritis |
| Pain NRS | weekly averages of daily pain numeric rating scale |
| P1NP | N-terminal propeptide of procollagen type I |
| PPAS | Per-Protocol Analysis Set |
| PPASB | Per-Protocol Analysis Set Phase B |
| qCT | quantitative computed tomography |
| RTSM | Randomization and Trial Supply Management |
| SAE | serious adverse event |


| Abbreviation | Term |
|---|---|
| SAP | statistical analysis plan |
| SAS | Safety Analysis Set |
| SASB | Safety Analysis Set Phase B |
| SD standard deviation | |
| SI International System of Units | |
| WOMAC | Western Ontario and McMaster Universities Osteoarthritis Index |
| WOMAC Function | WOMAC physical function subscore |
| WOMAC Pain | WOMAC pain subscore |


#### 1 BACKGROUND

Osteoarthritis (OA) is the most common form of arthritis and the major cause of activity limitation and physical disability in older people. Today, 35 million people (13% of the US population) are 65 and older, and more than half of them have radiological evidence of OA in at least one joint. By 2030, 20% of Americans (about 70 million people) will have passed their 65th birthday and will be at risk for OA (Nevitt, Felson, & Lester, 2006).

The exact cause of OA is unknown, but it is associated with aging and normal wear on a joint. OA is characterized by the destruction of the articular cartilage, subchondral bone alterations, and synovitis. Patients present with pain and stiffness in their joints, with joints becoming stiffer and more immobile over time (Dougados & Hochberg, 2011). OA is a leading cause of physical disability in the US (Lawrence, et al., 2008).

Non-pharmacological management of OA (e.g., education, exercise, weight reduction) can only slightly reduce symptoms in affected joints (Bannuru, Kent, & McAlindon, 2015) (McAlindon, et al., 2014). Pharmacological management, specifically nonsteroidal anti-inflammatory drug (NSAID) use, has limited impact on clinical outcomes (Bellamy, et al., 2015) (Lapane, et al., 2015). Moreover, any clinical effects are short-lived and the potential side effects (particularly of oral NSAIDs), including but not limited to, cardiac, renal, and gastrointestinal (GI) effects, limit long-term use. Opioids are also frequently used in the management of OA pain, but have numerous potential side effects, ranging from addiction, a major public health concern in the US, to increased risk of falls, especially in the elderly.

There is a significant unmet need for pharmacological agents with disease-modifying properties for the treatment of OA. Most current treatments are designed only to relieve pain and reduce or prevent the disability caused by bone and cartilage degeneration. Available drug therapies target the symptoms, but not the cause, of this disease and no treatment inhibits or reverses the degenerative structural changes that are responsible for its (Nevitt, Felson, & Lester, 2006). There is a need for pharmacological agents to treat OA that have disease-modifying properties, but can also provide symptom relief (decreased pain and improved function), while still being safe to use by patients with comorbid conditions or concomitant medications (Pham, et al., 2003). Such agents could also potentially delay or reduce the need for joint replacement surgery, an end-stage option which may not be suitable for OA patients in which surgical risk is deemed too high.

In order to address the need for effective pharmaceutical agents to treat OA, Samumed has used structure-based drug design to synthesize a small molecule inhibitor of the Wnt pathway, lorecivivint (LOR; previously SM04690), as a potential OA therapeutic to be administered as a local injection in the affected joint. The Wnt pathway plays a central role in the initiation and progression of OA pathology and is crucial in normal joint metabolism (Hochberg, et al., 2012). The Wnt pathway is a major regulator of joint development and is involved in the formation of bone, cartilage, and synovium. In osteoarthritic joints, increased Wnt signaling stimulates cartilage-destroying protease production and drives local progenitor cells to become bone-forming osteoblasts instead of cartilage-forming chondrocytes, thereby contributing to

osteophyte formation and cartilage loss (Gelse, et al., 2012). Gene polymorphisms involved in Wnt signaling are associated with an increased susceptibility to OA development (Wu, et al., 2012). Established research suggests that modulation of Wnt signaling is an attractive target for the treatment of OA.

Lorecivivint inhibits the Wnt pathway through the dual inhibition of intranuclear kinases CLK2 and DYRK1A, and thereby potentially (a) reduces signs and symptoms of knee OA via an anti-inflammatory mechanism, (b) inhibits cartilage breakdown through effects on degradative enzymes, and (c) enhances formation of cartilage through effects on progenitor cells and chondrocytes residing in the joint. Thus, LOR has the potential to affect both structural and symptomatic mechanisms underlying OA. In a previous randomized controlled, 52-week Phase 2a trial, LOR demonstrated significant improvements compared with placebo in pain, function, and medial joint space width (mJSW) in subjects with moderately to severely symptomatic knee OA (Yazici, et al., 2020). In clinical studies to date, LOR has been well tolerated with a safety profile similar to that of placebo.

#### 2 OVERVIEW

This study was a multicenter, randomized, double-blind, placebo-controlled, parallel group study of a single concentration of SM04690 injected every 6 months into the target knee joint of moderately to severely symptomatic OA subjects. In this study, "placebo" refers to vehicle.

#### 3 STUDY OBJECTIVES AND ENDPOINTS

# 3.1 Study Objective

#### 3.1.1 Primary Objective

The primary objective of this study was to evaluate the safety and tolerability of SM04690 Injectable Suspension administered every 6 months through 52 weeks for the treatment of knee osteoarthritis (OA).

#### 3.1.2 Secondary Objectives

The secondary objectives of this study were:

- 1. To evaluate the effectiveness of SM04690 Injectable Suspension administered every 6 months through 52 weeks for the treatment of knee OA
- 2. To evaluate the use of quantitative computed tomography (qCT) to assess knee bone mineral density (BMD)
- 3. To evaluate the safety, tolerability, and effectiveness of SM04690 Injectable Suspension from 52 weeks through 104 weeks

#### 3.2 Study Endpoints

#### 3.2.1 Phase A General Safety Endpoints

1. Adverse events (AEs), serious adverse events (SAEs), vital signs, and clinical laboratory measures through Week 52

#### 3.2.2 Phase A Bone Imaging Endpoints

- 1. Actual BMD and change from baseline in BMD in the target knee as assessed by qCT through Week 52 compared to placebo
- 2. Within-subject difference in BMD from baseline through Week 52 between the target and non-target knee by qCT for SM04690
- 3. Within-subject difference in BMD from baseline through Week 52 between the target and non-target knee by qCT for placebo
- 4. Change from baseline in BMD in the spine and hips as assessed by dual-energy X-ray absorptiometry (DXA) at Week 24 and 52

# 3.2.3 Phase A Efficacy Endpoints

- 1. Characterization of change in OA pain in the target knee as measured by the weekly averages of daily pain numeric rating scale (NRS) from baseline through Week 52 accounting for repeated injections
- 2. Characterization of change durability of treatment response in OA pain in the target knee as measured by the weekly averages of daily pain NRS through Week 52 elapsed from prior injection to repeat injection
- 3. Characterization of change in OA function in the target knee as measured by WOMAC physical function subscore (WOMAC Function) from baseline through Week 52 accounting for repeated injections
- 4. Characterization of change durability of treatment response in OA function in the target knee as measured by WOMAC Function through Week 52 elapsed from prior injection to repeat injection
- 5. Characterization of change in medial joint space width (mJSW) as measured by radiograph of the target knee from baseline through Week 52 accounting for repeated injections
- 6. Characterization of change durability of treatment response in mJSW as measured by radiograph of the target knee through Week 52 elapsed from prior injection to repeat injection
- 7. Characterization of change in OA pain in the target knee as measured by WOMAC pain subscore (WOMAC Pain) from baseline through Week 52 accounting for repeated injections
- 8. Characterization of change durability of treatment response in OA pain in the target knee as measured by WOMAC Pain through Week 52 elapsed from prior injection to repeat injection
- 9. Characterization of change in OA disease activity as measured by Patient Global Assessment from baseline through Week 52 accounting for repeated injections
- 10. Characterization of change durability of treatment response in OA disease activity as measured by Patient Global Assessment through Week 52 elapsed from prior injection

to repeat injection

#### 3.2.4 Phase A Exploratory Biomarker Endpoints

1. Change from baseline in serum bone biomarkers (e.g., N-terminal propeptide of procollagen type I [P1NP] and  $\beta$ -C-terminal telopeptide [ $\beta$ -CTX]) and a serum cartilage biomarker (e.g., cartilage oligomeric matrix protein [COMP]) through Week 52 compared to placebo

#### 3.2.5 Phase B General Safety Endpoints

1. AEs, SAEs, vital signs, and clinical laboratory measures from Week 52 through Week 104

# 3.2.6 Phase B Bone Imaging Endpoints

- 1. Actual BMD and change from baseline in BMD in the target knee as assessed by qCT through Week 104 compared to placebo
- 2. Within-subject difference in BMD from baseline through Week 104 between the target and non-target knee by qCT for SM04690
- 3. Within-subject difference in BMD from baseline through Week 104 between the target and non-target knee by qCT for placebo
- 4. Change from baseline in BMD in the spine and hips as assessed by DXA through Week 104

#### 3.2.7 Phase B Efficacy Endpoints

- 1. Characterization of change in OA pain in the target knee as measured by the weekly averages of daily pain NRS from baseline through Week 104 accounting for repeated injections
- 2. Characterization of change durability of treatment response in OA pain in the target knee as measured by the weekly averages of daily pain NRS through Week 104 elapsed from prior injection to repeat injection
- 3. Characterization of change in OA function in the target knee as measured by WOMAC Function from baseline through Week 104 accounting for repeated injections
- 4. Characterization of change durability of treatment response in OA function in the target knee as measured by WOMAC Function through Week 104 elapsed from prior injection to repeat injection
- 5. Characterization of change in mJSW as measured by radiograph of the target knee from baseline through Week 104 accounting for repeated injections
- 6. Characterization of change durability of treatment response in mJSW as measured by radiograph of the target knee through Week 104 elapsed from prior injection to repeat injection
- 7. Characterization of change in OA pain in the target knee as measured by WOMAC Pain from baseline through Week 104 accounting for repeated injections
- 8. Characterization of change durability of treatment response in OA pain in the target knee as measured by WOMAC Pain through Week 104 elapsed from prior injection to repeat injection
- 9. Characterization of change in OA disease activity as measured by Patient Global

Assessment from baseline through Week 104 accounting for repeated injections

10. Characterization of change durability of treatment response in OA disease activity as measured by Patient Global Assessment through Week 104 elapsed from prior injection to repeat injection

#### 3.2.8 Phase B Exploratory Biomarker Endpoints

1. Change from Week 52 in serum bone biomarkers (e.g., P1NP and β-CTX) and a serum cartilage biomarker (e.g., COMP) through Week 104

# 4 OVERALL STUDY DESIGN AND PLAN

This study was a multicenter, randomized, double-blind, placebo-controlled, parallel group study of a single concentration of SM04690 injected into the target knee joint of moderately to severely symptomatic OA subjects.

## **Core Phase (Phase A)**

Subjects participated in a screening period of a minimum of 10 days and up to 19 days and a 52-week evaluation period. Each subject was to receive an injection on Day 1 and Week 24 (same dose for each injection) and was to be observed for one year after first injection.

### **Extension Phase (Phase B)**

Subjects who completed Phase A were eligible to enter the extension phase, Phase B, for an additional 52 weeks of treatment. Subjects remained on their randomized treatment (SM04690 or placebo) for the additional year. Each subject was to receive an injection at Week 52 [Phase A End of Study (EOSa)] and Week 76.

#### 4.1 Selection of Study Population

The study population included ambulatory males and females between 40 and 80 years of age, inclusive, with moderately to severely symptomatic knee OA. Complete inclusion/exclusion criteria are available in the study protocol.

#### 4.2 Method of Treatment Assignment and Randomization

Approximately 100 subjects were randomized 1:1 to one of two treatment groups (0.07 mg active per 2 mL injection : 2 mL placebo) using a permuted block design via Medidata Rave Randomization and Trial Supply Management (RTSM). Fifty blocks of size 4 were generated for a total of 200 possible subject slots.

# 4.3 Treatment Blinding

Phase A of the study was double-blind. Study medication was provided to the investigational center, and the center identified unblinded personnel who were able to prepare and perform the injection of study medication and/or placebo. Study personnel administering or preparing study medication and reference therapy were to minimize any contact with the subject following the injection and not perform any study assessments throughout the duration of the study. Each site was required to document a blinding plan that identified the blinded and unblinded personnel at the investigational center and described how the study blind will be maintained.


Primary analysis of Phase A data was completed after the last subject completed Week 52 (EOSa). While the Sponsor was unblinded to study treatment after the Phase A analysis (after the last subject completed Week 52 [EOSa]), the Investigators and the subjects remained blinded for Phase B.

# 4.4 Minimization of Missing Data

#### 4.4.1 Collection of Clinical Outcomes

Clinical outcomes data were collected using electronic diary (see Protocol Section 7.3.8 for schedule of diary data collection). Eligibility criteria for the trial included successful completion of the electronic diary in the collection of both Pain NRS and WOMAC (see Inclusion Criteria 6-10). Use of electronic diary as well as enriching for subjects compliant with electronic diary use during the screening period were specific protocol strategies designed to minimize the loss of key endpoint data.

#### 4.4.2 Prohibited Medications, Treatments, and Procedures

During the conduct of the study, several medications, treatments, and procedures were prohibited (see Protocol Section 7.6). The overall intent of these prohibitions was to minimize any possible bias in the assessment of the clinical trial endpoints. However, the protocol did allow for the use of these prohibited therapies if and only if there were required to ensure subject safety. Investigators were instructed to notify the sponsor's Medical Monitor, who would note the prohibited therapy as a protocol deviation. Subjects were not automatically discontinued based upon prohibited therapy use, allowing for continued data collection and assessment of the impact of prohibited therapy on key endpoint data.

#### 4.4.3 Intermittent Missing Data

Ongoing programmatic surveillance of electronic diary and visit compliance using intranet dashboards during trial conduct led to the identification of subjects that were not compliant with their electronic diary entries. Sites were notified of possible non-compliant subjects and were instructed to address any possible technical or conduct issues with these subjects prior to key endpoint data collection times. The ongoing monitoring of electronic diary compliance was a specific strategy designed to minimize the loss of key endpoint data.

# 5 ANALYSIS AND REPORTING

#### 5.1 Phase A Analysis

Primary analysis of Phase A data was completed after the last subject completed the Week 52 (EOSa) visit. A separate SAP was prepared for Phase A analyses.

#### 5.2 Phase B Analysis

Phase B endpoints will be analyzed in a similar fashion as Phase A endpoints. This analysis plan is only focused on Phase B analysis.

#### 6 SAMPLE SIZE DETERMINATION

The sample size for this trial was based upon accepted investigational studies exploring changes in bone density.


Based upon the subchondral BMD data obtained using qCT in SM04690-01, a coefficient of variation (CV) of 0.30 was presumed to be shared by both treatment and placebo groups; this presumed CV is larger than the observed CVs in SM04690-01. Assuming a Type 1 error of 0.05, 100 subjects (50 subjects per group) will provide 81.6% power to estimate a BMD ratio (SM04690: placebo) of 0.93 with a one-sided confidence interval extending to 0.80 assuming a non-inferiority design.

## 7 ANALYSIS POPULATIONS

# 7.1 Full Analysis Set

The Full Analysis Set (FAS) includes all subjects who were randomized and received at least one study injection. The FAS is used to describe the analysis set which is as complete as possible and as close as possible to the intent-to-treat ideal of including all randomized subjects. Subjects will be analyzed as randomized for the FAS.

# 7.2 Full Analysis Set Phase B

The Full Analysis Set Phase B (FASB) includes all FAS subjects who received at least one study injection in Phase B. Subjects will be analyzed as randomized for the FASB.

#### 7.3 Modified Full Analysis Set

The modified Full Analysis Set (mFAS) includes all FAS subjects who received both scheduled Phase A injections into the target knee (Day 1, Week 24). Subjects will be analyzed as randomized for the mFAS.

# 7.4 Per-Protocol Analysis Set

The Per-Protocol Analysis Set (PPAS) includes all mFAS subjects who completed Phase A of the study (i.e. subjects who terminate the study early will be excluded) and did not have any protocol deviations that may have impacted the evaluation of efficacy outcomes (see Section 9.2). Subjects will be analyzed as randomized for the PPAS. A list of subjects excluded from PPAS can be found in the Phase A SAP.

#### 7.5 Per-Protocol Analysis Set Phase B

The Per-Protocol Analysis Set Phase B (PPASB) includes all PPAS who completed Phase B of the study and did not have any protocol deviations in Phase B that may have impacted the evaluation of efficacy outcomes (see Section 9.2). Subjects excluded from per-protocol analysis in Phase A are by definition excluded from per-protocol analysis in Phase B. Subjects will be analyzed as randomized for the PPASB.

#### 7.6 Safety Analysis Set

The Safety Analysis Set (SAS) includes all subjects who received at least one study injection. Subjects will be analyzed as treated on Day 1 for the SAS. In this study, the FAS and SAS are identical, but for consistency with other studies, the SAS will be used in summaries of safety.

#### 7.7 Safety Analysis Set Phase B

The Safety Analysis Set Phase B (SASB) includes all subjects who received at least one study injection in Phase B. Subjects will be analyzed as treated on Day 1 for the SASB. In this study,

the FASB and SASB are identical, but for consistency with other studies, the SASB will be used in summaries of safety.

# 8 GENERAL ISSUES FOR STATISTICAL ANALYSIS

#### 8.1 General Statistical Methodology

For continuous variables, the outcome measure at each visit, as well as the absolute change (outcome at visit – outcome at baseline), will be summarized within each treatment group using descriptive statistics (number of subjects, mean, standard deviation (SD), median, minimum, and maximum). The number of evaluable subjects in any analysis set may vary by endpoint/timepoint based on missing data. Categorical variables will be summarized with frequency tables.

All subject-level listings will be comprehensive and include subjects enrolled in both Phase A and Phase B. Data collected from unscheduled visits will not be included in summary tables but will be included in subject-level listings as appropriate.

#### 8.1.1 Baseline

Baseline is defined as the last value recorded for any given parameter prior to first study medication injection on Day 1. For qCT and DXA, values recorded from Screening Visit 2 will serve as baseline, regardless of whether the scans took place before or after first study medication injection. Baseline values for Phase B of the study are the same as they were for Phase A.

#### 8.1.2 Analysis of Covariance (ANCOVA)

ANCOVA models will be used to analyze change over time in bone imaging endpoints. All models will be adjusted for baseline. Least squares estimates, two-sided 95% confidence intervals (unadjusted for multiplicity), and effect sizes will be provided.

#### 8.1.3 Mixed-Effects Models for Repeated Measures

A mixed-effects model for repeated measures (MMRM) will be used to analyze change over time in Pain NRS. The model will be estimated assuming a Toeplitz variance-covariance matrix. The Toeplitz structure is a more generalized form of autogressive-1 (AR1) structure, allowing the data to inform how the correlation between within-subject observations decreases over time instead of implicitly defining a uniform decay structure (Kincaid, 2005).

MMRM presumes that missing data are not caused by something observable within the conduct of the trial (i.e. missing-at-random [MAR]). It is plausible to presume a MAR mechanism as there have been no observed tolerability issues to the administration of study injection during the prior development trials. Additionally, the study injection cannot be removed after it has been administered, eliminating study drug discontinuation as a source of treatment estimate confounding.


#### 8.1.4 Data Handling for Subjects Who Withdrew from Study

If a subject discontinues the study, early termination assessments will be performed according to the protocol. If these assessments occur during a scheduled visit, they will be associated with that visit for the purposes of analysis.

#### 8.1.5 Imputation of Missing Data

No imputation will be performed for Phase B efficacy analysis.

#### 8.2 General Safety Assessments

#### 8.2.1 Adverse Events

An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP or other protocol-imposed intervention, regardless of attribution. Signs and symptoms of exacerbation or worsening of target knee OA were captured in the context of efficacy assessments. Anticipated fluctuations or anticipated deterioration (in the opinion of the Investigator) of the underlying disease (target knee OA) were not considered as AEs.

Severity was assessed utilizing the CDISC AESEV, which classifies AEs as mild, moderate, or severe. For analysis, relationship will be dichotomized into Unrelated (combining Not Related and Unlikely Related) and Related (combining Possibly Related and Probably Related).

#### 8.2.2 Vital Signs and Weight

Vital signs were measured by a qualified staff member at all visits except Screening Visit 2. At each time point, the following vital signs were to be measured:

- Body temperature
- Pulse rate
- Respiratory rate
- Blood pressure (systolic and diastolic) after the subject rests (sitting or supine) for at least 5 minutes

Any measurement that was, in the opinion of the Investigator, abnormal AND clinically significant was considered as medical history if found prior to study medication injection or as an AE if found after study medication injection.

Weight measurements were to be taken at Screening Visit 1 and at Weeks 24, 52 (EOSa), 76, and 104 [Phase B End of Study (EOSb)] or ET.

#### 8.2.3 Clinical Laboratory Evaluations

Fasting samples for clinical laboratory analysis were to be collected at Screening Visit 2 and Weeks 4, 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb) or ET. At a minimum, the following tests were conducted:

• *Chemistry panel*: Albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, bicarbonate, calcium (corrected total), chloride, creatinine, glucose, lactate dehydrogenase, potassium, sodium, bilirubin (total)

- *Hematology*: Hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, and platelet count
- *Urinalysis:* Clarity, specific gravity, pH, protein, glucose, ketones, nitrite, leukocytes, and occult blood

Urine microscopy was to be performed if urinalysis urine protein, leukocyte esterase, occult blood, or nitrite values were out of range, or if the Investigator deemed that the microscopy was clinically warranted

# 8.3 Bone Imaging Assessments

#### 8.3.1 Knee BMD (qCT)

qCT scans of both knee joints were to be taken at Screening Visit 2 and at Weeks 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb) or ET. The qCT scans assessed changes in BMD in both tibias across three compartments (medial, lateral, and total [medial + lateral]) and four volumes of interest (subchondral epiphysis, mid-epiphysis, juxtaphysis, and total).

For analysis, values of BMD that have undergone longitudinal correction will be used when available. Refer to Bioclinica's *Imaging Review Charter* for details on how corrections may have been made for scanner quality control.

#### 8.3.2 Spine and Hip BMD (DXA)

Bone density DXA scans of the spine and hips were to be taken at Screening Visit 2 and at Weeks 24, 52 (EOSa), 76, and 104 (EOSb) or ET. Spine DXA scans assessed changes in BMD in two regions of interest: total (lumbar vertebrae L1 to L4) and adjusted total (L1 to L4 excluding any vertebral levels due to artifact). Hip DXA scans assessed changes in BMD in two regions of interest: total hip and femoral neck.

The DXA scanning assessed changes in the hips and spine and included the following parameters:

- BMD: individual subject's test, measured in g/cm<sup>2</sup>
- **T-score**: The number of standard deviations a subject's BMD differs from the mean BMD of a young, healthy sex-matched adult population
- **Z-score**: The number of standard deviations a subject's BMD differs from the mean BMD for an age-matched and sex-matched healthy population.

Negative T- and Z-scores indicate results below population mean, and positive scores indicate results above population mean. All T-scores were determined using reference data for Whites regardless of the individual subject's race. Z-scores were determined using African American reference data for Black or African American subjects. All other races or those with unknown race used the White reference data for Z-score calculations. Spine reference values were based on manufacturer's reference data; total hip reference values were based on NHANES-98 data.

For safety analysis, values of BMD and T-scores that have undergone longitudinal correction will be used when available. Refer to Bioclinica's *Imaging Review Charter* for details on how corrections may have been made for scanner quality control. Z-scores will not be summarized.


#### 8.4 Efficacy Assessments

#### 8.4.1 Pain NRS

The Pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the previous 24 hours, where 0 represents no pain and 10 represents extreme pain. Subjects were prompted on their electronic device to report average pain daily (between 5:00 pm and 11:59 pm) in both knees at Screening Visit 2 and on the target knee only through the end of the study. An average weekly score (referred to as Pain NRS) will be calculated for each subject if they had provided a response for at least 4 out of 7 days in a given week. Weeks are defined as Day -7 through Day -1 (day before treatment) for baseline, Day 1 (day of treatment) through Day 7 for Week 1, Day 8 through Day 14 for Week 2, and so on as detailed in Appendix 1. The day on which subjects completed their scheduled study visits (e.g. Week 4 Visit, Week 12 Visit, etc.) does not impact the above definition of weeks.

#### 8.4.2 WOMAC

The WOMAC is a widely used, proprietary outcome measurement tool used by health professionals to evaluate the condition of patients with OA of the knee and hip, including pain, stiffness, and physical functioning of a target joint. The WOMAC Version NRS 3.1 questionnaire were to be completed by the subject for their target knee in the evening (between 5:00 pm and 11:59 pm) remotely on their electronic device 5 days after Screening Visit 2 or up until the day before the Day 1 visit. After Day 1, monthly (every 4 weeks, with a window of  $\pm$  3 days) WOMAC assessments were to be completed by the subjects for their target knee in the evening (between 5:00 pm and 11:59 pm) remotely on their electronic devices. At Weeks 24, 52 (EOSa), and 76, the WOMAC questionnaire must have been completed prior to the study medication injection; otherwise the results were not used in analysis. If an assessment was completed more than once within a window, only the first assessment will be used for analysis. All visit windows are detailed in Appendix 1.

WOMAC consists of 24 questions in three domains: physical function (17 questions), pain (5 questions) and stiffness (2 questions). The response for each question in the NRS format ranges from 0 to 10. Each domain subscore as well as a total score are calculated by adding together the numerical responses for a range of 0 to 240 total points. For analysis, WOMAC scores will be linearly transformed to a 0-100 scale, where 0 represents no difficulty and 100 represents extreme difficulty.

#### 8.4.3 Patient Global Assessment of Disease Activity

The Patient Global Assessment is an 11-point [0-10] NRS on which the subjects rated how they felt their target knee OA was, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right). The Patient Global Assessments were to be completed by the subject in the evening (between 5:00 pm and 11:59 pm) remotely on their electronic device 5 days after their Screening Visit 2 or up until the day before the Day 1 visit. After Day 1, monthly (every 4 weeks, with a window of  $\pm$  3 days) Patient Global Assessments were to be completed by the subjects in the evening (between 5:00 pm and 11:59 pm) remotely on their electronic devices. At Weeks 24, 52 (EOSa), and 76, the Patient Global Assessment must have been completed prior to the study

medication injection; otherwise the results were not used in analysis. If an assessment was completed more than once within a window, only the first assessment will be used for analysis. All visit windows are detailed in Appendix 1.

For analysis, scores will be linearly transformed to a 0-100 scale, where 0 represents "Very Good" and 100 represents "Very Bad". If an assessment was completed more than once within a window, only the first assessment will be used for analysis.

#### 8.4.4 mJSW

Radiographs of the knee joints were to be taken at Screening Visit 1 and at Weeks 24, 52 (EOSa), 76, and 104 (EOSb) or ET. Bilateral radiographs were to be taken in a weight-bearing fixed flexion position, using a posterior-anterior view X-ray. All radiographs were submitted to an independent radiologist at the central imaging vendor who documented disease stage according to the Kellgren-Lawrence grading scale for compliance with inclusion/exclusion criteria, as well as mJSW for efficacy assessments. mJSW measurements will be reported to two decimal places.

#### 8.5 Exploratory Biomarker Assessments

Blood samples for biomarker analysis were to be collected at Screening Visit 2 and Weeks 4, 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb) or ET. Biomarkers that were assessed included, but were not limited to, bone biomarkers (P1NP and β-CTX) and a cartilage biomarker (COMP).

## 9 STUDY SUBJECTS AND DEMOGRAPHICS

# 9.1 Disposition of Subjects and Withdrawals

Subject disposition will be presented in a summary table detailing the number and percentage of subjects who were randomized, treated in Phase B, completed Phases A and B of the study, and discontinued (e.g. subject withdrawal, adverse event, etc.) overall and by treatment group. Additionally, subject disposition for randomized subjects will be presented by treatment group and study site. Additional tables will be prepared to summarize the number of subjects enrolled under each protocol version and included in each Phase B analysis set. The disposition for individual subjects will be listed along with additional information on discontinued subjects.

#### 9.2 Protocol Deviations

A protocol deviation is defined as any noncompliance with the clinical trial protocol requirements. The noncompliance may be either on the part of the subject, the Investigator, or the study site staff.

Deviations are summarized into one of the following categories:

- Investigational Product
- Informed Consent
- Enrollment
- Procedures
- Labs/Specimens
- Study Visits
- Source Documentation


- Diaries, Questionnaires, or Patient Reported Outcomes
- Subject Non-Compliance
- Serious Adverse Events

Deviations are categorized as major or minor by a cross-functional team according to pre-defined criteria established in the Protocol Deviation Classification Guideline.

- A major deviation is defined as a divergence from the protocol that materially (a) reduces the quality or completeness of efficacy data, (b) makes the informed consent inaccurate, or (c) impacts a subject's safety, rights or welfare.
- A minor deviation is defined as a divergence from the protocol that deviates from the
  procedures and guidelines outlined in the protocol, but is not classified as a major
  deviation (i.e. the deviation does not materially (a) reduce the quality or completeness of
  the data, (b) make the informed consent inaccurate, or (c) impact a subject's safety, rights
  or welfare).

Protocol deviations may result in subject exclusion from the PPASB. Prior to Phase B database lock, all protocol deviations were reviewed by study team members to determine if the deviation could reasonably affect/confound interpretation of efficacy endpoints and should result in the subject being excluded from the PPASB. Subjects with the following types of deviations were excluded from the PPASB:

• Subjects taking pain medications that may significantly impact pain and function assessment

A final list of protocol deviations resulting in subject exclusion from the PPAS and PPASB can be found in Appendix 2.

Major protocol deviations that occurred in Phase B will be summarized by site and category, and all protocol deviations will be listed for each subject. Additionally, the COVID-19 pandemic related protocol deviations that occurred in Phase B will be summarized separately.

For deviations associated with a study visit, only those occurring at Week 64, Week 76, Week 88, or Week 104 (EOSb) will count as Phase B deviations. For deviations not associated with a study visit (e.g. prohibited medications), the dates listed in the CRA comments were evaluated against the date of the subject's Week 52 injection. Any deviations that occurred after the Week 52 injection will be counted as Phase B deviations. Details can be found in Appendix 3.

# 9.3 Demographics and Other Baseline Characteristics

Demographic and baseline characteristics of subjects in Phase B, including sex, race, ethnicity, age at baseline, weight, height, body mass index, KL grade, WPI, SSQ2, and mJSW, will be presented overall and by treatment group. Continuous variables will be summarized with descriptive statistics and categorical variables will be summarized with frequencies and percentages. The summaries will be provided for the FASB and PPASB. Subject-level listings will be provided.


#### 9.4 Medical History

A summary of medical history by MedDRA system organ class was provided in the Phase A analysis. A subject-level listing will provide further information on each event.

#### 10 GENERAL SAFETY ANALYSIS

Whereas Phase A analysis (defined prior to unblinding) was the primary analysis for this study, data collected during Phase B complements the primary analysis by offering insight into safety after more than one year of treatment.

#### 10.1 Adverse Events

AEs collected in this study are events that occur during the course of the study that are not present prior to Day 1 study medication injection, or, if present at the time of study medication injection, have worsened in severity during the course of the study. AEs will be presented in summary tables depicting the number and percent of unique subjects experiencing each AE and the number of AEs overall and within each treatment group. The following summaries will be provided for both the entire study length (SAS) and for Phase B (SASB) separately:

- All AEs by seriousness, severity, and relationship to study product
- AEs by highest degree of seriousness, severity, and relationship to study drug
- AEs by MedDRA system organ class and preferred term
- AEs and SAEs by preferred term incidence
- Target-knee-related AEs and SAEs by preferred term incidence
- SAEs in subjects diagnosed with COVID-19

Subject-level listings will be provided for all AEs and all SAEs separately.

#### 10.2 Vital Signs and Weight

Weight and vital signs (including systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, and body temperature) will be summarized for each treatment group. A comprehensive statistical description (number of subjects, mean, standard deviation, median, minimum, and maximum) of each parameter at baseline will be provided along with the change from baseline at each subsequent visit for subjects in the SAS. A subject-level listing will be provided.

# 10.3 Clinical Laboratory Evaluations

All chemistry, hematology and urinalysis results from the central laboratory will be comprehensively summarized into shift tables as normal, non-clinically significant abnormal, and clinically significant abnormal. Assessments of clinical significance for abnormal values were made by the investigator on results that were outside of the normal range. Comprehensive shift tables will compare the number and percent of assessments from each visit to baseline values for each treatment group.

All chemistry and hematology results from the central laboratory will be comprehensively summarized for each treatment group. Descriptive statistics of each laboratory test at all


timepoints will be provided along with the change from baseline at each subsequent timepoint for subjects in the SAS. The International System of Units (SI) will be used for all summaries.

Abnormal chemistry, hematology, urinalysis, and urine microscopy results for each subject will be provided in listings that will include laboratory test name, result, normal range, and an explanation for clinically significant values.

#### 11 BONE IMAGING ANALYSIS

Whereas Phase A analysis (defined prior to unblinding) was the primary analysis for this study, data collected during Phase B complements the primary analysis by offering insight into safety after more than one year of treatment. Bone imaging analysis will be performed on the SAS.

A statistical description of target knee, non-target knee, spine, and hip BMD at baseline will be provided along with absolute and percent changes from baseline at each subsequent timepoint. Statistical descriptions of knee BMD for subgroups such as KL grade, sex, and age group may be provided.

Difference between target knee and non-target knee BMD will be summarized at baseline along with absolute changes from baseline at each subsequent timepoint. Spine and Hip BMD T-scores will be summarized at baseline only for subjects enrolled in Phase B.

Baseline-adjusted ANCOVA as described in Section 8.1.2 will be used to analyze the change from baseline in BMD in the target knee and evaluated at Weeks 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb).

Baseline-adjusted ANCOVA will also be used to analyze the within-subject difference in BMD between the target and non-target knee by qCT for SM04690, within-subject difference in BMD between the target and non-target knee by qCT for placebo, and change from baseline in BMD of the spine and hips by DXA for SM04690 subjects versus placebo. The models will be evaluated at Weeks 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb) for qCT and Weeks 24, 52, 76, and 104 (EOSb) for DXA.

Knee BMD analysis will include all compartments and volumes of interest. Spine BMD analysis will include the adjusted total region of interest; hip BMD analysis will include both total hip and femoral neck regions of interest.

Subject-level listings will be provided.

#### 12 EFFICACY ANALYSIS

A statistical description of Pain NRS at baseline will be provided along with absolute changes from baseline at each subsequent timepoint for subjects in the FASB and PPASB. Statistical descriptions of WOMAC Pain, WOMAC Function, Patient Global Assessment, and mJSW at baseline will also be provided along with absolute changes from baseline at each subsequent timepoint for subjects in the FASB only.


Changes in the target knee from baseline in Pain NRS will be characterized using MMRM for subjects in the FASB and PPASB; the models will be evaluated through Week 104 (EOSb). All models will use treatment group, week, treatment×week interaction, and baseline values as covariates. Unadjusted 95% confidence intervals and P values will be reported.

If a subject submitted data related to their non-target knee due to an electronic device error, this data will not be analyzed.

Subject-level listings will be provided.

Since Phase A analysis (defined prior to unblinding) was the primary analysis for this study, there will be no estimands provided for Phase B.

# 13 EXPLORATORY BIOMARKER ANALYSIS

A statistical description of biomarkers COMP, P1NP, and  $\beta$ -CTX at baseline will be provided along with absolute and percent changes from baseline at each subsequent timepoint for subjects in the SAS.

Baseline-adjusted ANCOVA will also be used to analyze the change from baseline in these biomarkers and evaluated at Weeks 4, 12, 24, 36, 52 (EOSa), 64, 76, 88, and 104 (EOSb). Subject level listings will be provided.

#### 14 MEDICATIONS

The summary of medications will be performed on the SASB.

#### 14.1 Concomitant Medications

The World Health Organization Drug Dictionary (WHODD) will be used to classify prior and concomitant medications by Anatomical Main Group (Anatomical Therapeutic Chemical, ATC, Level 1), Therapeutic Subgroup (ATC Level 2), and preferred term. Prior and concomitant medication usage will be summarized by the number and percentage of subjects receiving each medication by treatment group.

The subgroup of medications initiated after Week 52 injection will be summarized in the same manner. If a medication start date is incomplete, it will be imputed with the latest possible date to increase the likelihood it is included in the table of medications initiated after first exposure. For example, medication start dates of "2019" and "2020-02" would be imputed to "2019-12-31" and "2020-02-29", respectively.

Subject-level listings containing prior and concomitant medications (WHODD coding), and procedures/non-drug therapies (MedDRA coding) will be provided and will display the dates as they were entered (not the imputed version described above).

#### 14.2 Exposure

All treated subjects were scheduled to receive two injections during Phase A of the trial and two injections during Phase B of the trial. A summary table of the number injections received will be provided. A list of lot numbers used in this study will be provided in the clinical study report.

# 15 CHANGES TO PLANNED ANALYSIS

For the Phase B exploratory biomarker endpoint, all changes were calculated from baseline instead of from Week 52.

# 16 REFERENCES

- Bannuru, R. R., Kent, D. M., & McAlindon, T. E. (2015, May 5). Pharmacologic Interventions for Knee Osteoarthritis. *Annals of Internal Medicine*, 162(9), 672. doi:10.7326/L15-5090-2.
- Bellamy, N., Hochberg, M., Tubach, F., Martin-Mola, E., Awada, H., Bombardier, C., . . . Dougados, M. (2015, Jul 6). Development of multinational definitions of minimal clinically important improvement and patient acceptable symptomatic state in osteoarthritis. *Arthritis Care & Research*, 67(7), 972-80. doi:10.1002/acr.22538
- Dougados, M., & Hochberg, M. C. (2011). Management of osteoarthritis. In M. C. Hochberg, A. J. Silman, M. E. Smolen, M. E. Weinblatt, & M. H. Weisman, *Rheumatology*. Elsevier, PA.
- Gelse, K., Ekici, A. B., Cipa, F., Swoboda, B., Carl, H. D., Olk, A., . . . Klinger, P. (2012, Feb). Molecular differentiation between osteophytic and articular cartilage--clues for a transient and permanent chondrocyte phenotype. *Osteoarthritis Cartilage*, 20(2), 162-71. doi:10.1016/j.joca.2011.12.004
- Hochberg, M. C., Altman, R. D., April, K. T., Benkhalti, M., Guyatt, G., Mcgowan, J., . . . Tugwell, P. (2012, Apr). American College of Rhemuatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. *Arthritis Care & Research*, 64(4), 465-474. doi:10.1002/acr.21596
- Kincaid, C. D. (2005). Guidelines for Selecting the Covariance Structure in Mixed Model Analysis. *Proceedings of the Thirtieth Annual SAS Users Group International Conference*.
- Lapane, K. L., Yang, S., Driban, J. B., Liu, S. H., Dube, C. E., McAlindon, T. E., & Eaton, C. B. (2015, Nov 4). Effects of prescription nonsteriodal antiinflammatory drugs on symptoms and disease progression among patients with knee osteoarthritis. *Arthritis & Rheumatology*, 67(3), 724-32. doi:10.1002/art.38933
- Lawrence, R. C., Felson, D. T., Helmick, C. G., Arnold, L. M., Choi, H., Deyo, R. A., . . . Wolfe, F. (2008). Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. *Arthritis & Rheumatology*, 58(1), 26-35. doi:10.1002/art.23176
- McAlindon, T. E., Bannuru, R. R., Sullivan, M. C., Arden, N. K., Berenbaum, F., Bierma-Zeinstra, S. M., . . . Underwood, M. (2014, Mar). OARSI guidelines for the non-surgical management of knee osteoarthritis. *Osteoarthritis Cartilage*, 22(3), 363-88. doi:10.1016/j.joca.2014.01.003

- Nevitt, M. C., Felson, D. T., & Lester, G. (2006, Jun 21). *Osteoarthritis Initiative: A Knee Health Study*. Retrieved from OARSI Journal: https://www.oarsijournal.com/cms/10.1016/j.joca.2016.09.013/attachment/17129285-04bf-4f1c-a2f4-6c3f498da638/mmc2.pdf
- Pham, T., Van Der Heijde, D., Lassere, M., Altman, R. D., Anderson, J. J., Bellamy, N., . . . Dougados, M. (2003, Jul). Outcome variables for osteoarthritis clinical trials: The OMERACT-OARSI set of responder criteria. *Journal of Rheumatology*, 30(7), 1648-54.
- Wu, L., Huang, X., Li, L., Huang, H., Xu, R., & Luyten, W. (2012). Insights on biology and pathology of HIF-1α/-2α, TGFβ/BMP, Wnt/β-catenin, and NF-κB pathways in osteoarthritis. *Current Pharmaceutical Design*, *18*(22), 3293-312. doi:10.2174/1381612811209023293
- Yazici, Y., McAlindon, T. E., Gibofsky, A., Lane, N. E., Clauw, D., Jones, M., . . . Hochberg, M. C. (2020, Oct). Lorecivivint, a Novel Intraarticular CDC-like Kinase 2 and Dual-Specificity Tyrosine Phosphorylation-Regulated Kinase 1A Inhibitor and Wnt Pathway Modulator for the Treatment of Knee Osteoarthritis: A Phase II Randomized Trial. *Arthritis & Rheumatology*, 72(10), 1694-1706. doi:10.1002/art.41315

# 17 APPENDICES

# 17.1 Appendix 1 – Visit Windows

| Baseline Last value before first injection Week 1 Image: square process of the | Pain NRS Day -7 to -1 Day 1 to 7 Day 8 to 14 Day 15 to 21 Day 22 to 28 Day 29 to 35 Day 26 to 42 Day 43 to 49 Day 50 to 56 Day 57 to 63 Day 64 to 70 |
|---|---|
| Week 1 Jean Strain | Day 1 to 7 Day 8 to 14 Day 15 to 21 Day 22 to 28 Day 29 to 35 Day 26 to 42 Day 43 to 49 Day 50 to 56 Day 57 to 63 |
| Week 2 I Week 3 Day 26 to 32 Week 4 Day 26 to 32 Week 5 D Week 6 D Week 7 D Week 8 Day 54 to 60 Week 9 D Week 10 D Week 11 D Week 12 Day 82 to 88 Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 D Week 17 D Week 18 D D Week 19 D D Week 20 Day 138 to 144 D Week 21 D D Week 22 D D | Day 8 to 14 Day 15 to 21 Day 22 to 28 Day 29 to 35 Day 26 to 42 Day 43 to 49 Day 50 to 56 Day 57 to 63 |
| Week 3 Day 26 to 32 Day 26 to 32 Week 5 Day 26 to 32 Day 26 to 32 Week 6 Day 54 to 60 Day 54 to 60 Week 8 Day 54 to 60 Day 54 to 60 Week 10 Day 54 to 60 Day 54 to 60 Week 10 Day 54 to 60 Day 54 to 60 Week 11 Day 82 to 88 Day 62 Week 12 Day 82 to 88 Day 62 Week 13 Day 62 Day 62 Week 14 Day 70 Day 70 Week 15 Day 70 Day 70 Week 16 Day 110 to 116 Day 70 Week 18 Day 70 Day 70 Week 20 Day 138 to 144 Day 70 Week 21 Day 70 Day 70 Week 22 Day 70 Day 70 Week 23 Day 70 Day 70 | Pay 15 to 21 Pay 22 to 28 Pay 29 to 35 Pay 26 to 42 Pay 43 to 49 Pay 50 to 56 Pay 57 to 63 |
| Week 4 Day 26 to 32 D Week 5 D Week 6 D Week 7 D Week 8 Day 54 to 60 Week 9 D Week 10 D Week 11 D Week 12 Day 82 to 88 Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 22 to 28 Pay 29 to 35 Pay 26 to 42 Pay 43 to 49 Pay 50 to 56 Pay 57 to 63 |
| Week 5 D Week 6 D Week 7 D Week 8 Day 54 to 60 D Week 9 D Week 10 D Week 11 D Week 12 Day 82 to 88 D Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 29 to 35 Pay 26 to 42 Pay 43 to 49 Pay 50 to 56 Pay 57 to 63 |
| Week 6 Day 54 to 60 Day 54 to 60 Week 8 Day 54 to 60 Day 54 to 60 Week 9 Day 54 to 60 Day 54 to 60 Week 10 Day 54 to 60 Day 54 to 60 Week 10 Day 54 to 60 Day 54 to 60 Week 11 Day 54 to 60 Day 54 to 60 Week 12 Day 82 to 88 Day 54 to 88 Week 13 Day 62 to 88 Day 62 to 88 Week 14 Day 62 to 88 Day 62 to 88 Day 62 to 88 Week 14 Day 75 to | Pay 26 to 42 Pay 43 to 49 Pay 50 to 56 Pay 57 to 63 |
| Week 8 Day 54 to 60 Day 54 to 60 Week 9 Day 54 to 60 Day 54 to 60 Week 10 Day 62 to 80 Day 62 Week 11 Day 82 to 88 Day 62 Week 12 Day 82 to 88 Day 62 Week 13 Day 62 Day 62 Week 14 Day 62 Day 62 Week 15 Day 62 Day 62 Week 15 Day 62 Day 62 Week 16 Day 110 to 116 Day 62 Week 17 Day 62 Day 62 Week 18 Day 710 to 116 Day 710 to 116 Week 19 Day 710 to 116 Day 710 to 116 Week 20 Day 138 to 144 Day 710 to 116 Week 21 Day 710 to 116 Day 710 to 116 Week 22 Day 710 to 116 Day 710 to 116 | Pay 43 to 49 Pay 50 to 56 Pay 57 to 63 |
| Week 8 Day 54 to 60 D Week 9 D D Week 10 D D Week 11 D D Week 12 Day 82 to 88 D Week 13 D D Week 14 D D Week 15 Day 110 to 116 Da Week 16 Day 110 to 116 Da Week 17 Da Da Week 18 Da Da Week 19 Da Da Week 20 Day 138 to 144 Da Week 21 Da Da Week 22 Da Da Week 23 Da Da | Pay 50 to 56 Pay 57 to 63 |
| Week 9 D Week 10 D Week 11 D Week 12 Day 82 to 88 Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 57 to 63 |
| Week 10 D Week 11 D Week 12 Day 82 to 88 Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Week 21 Da Week 22 Da Week 23 Da | • |
| Week 12 Day 82 to 88 D Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Week 21 Da Week 22 Da Week 23 Da | Pay 64 to 70 |
| Week 12 Day 82 to 88 D Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | ay of to 70 |
| Week 13 D Week 14 D Week 15 D Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 71 to 77 |
| Week 14 Day Week 15 Day Week 16 Day 110 to 116 Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 78 to 84 |
| Week 15 Day 110 to 116 Da Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 85 to 91 |
| Week 16 Day 110 to 116 Da Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | Pay 92 to 98 |
| Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | ay 99 to 105 |
| Week 17 Da Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | y 106 to 112 |
| Week 18 Da Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | y 113 to 119 |
| Week 19 Da Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | y 120 to 126 |
| Week 20 Day 138 to 144 Da Week 21 Da Week 22 Da Week 23 Da | xy 127 to 133 |
| Week 21 Da Week 22 Da Week 23 Da | y 134 to 140 |
| Week 22 Da Week 23 Da | y 141 to 147 |
| Week 23 Da | y 148 to 154 |
| | y 155 to 161 |
| | y 162 to 168 |
| · | y 169 to 175 |
| | y 176 to 182 |
| | y 183 to 189 |
| | y 190 to 196 |
| · | y 197 to 203 |
| | xy 204 to 210 |
| | y 211 to 217 |
| | xy 218 to 224 |
| , and the second | • |
| | v 225 to 231 |
| | y 225 to 231<br>y 232 to 238 |
| | y 232 to 238 |
| Week 37 Day 230 to 230 Day | • |

| Week 38 | | Day 260 to 266 |
|----------------|-----------------|----------------|
| Week 39 | | Day 267 to 273 |
| Week 40 | Day 278 to 284 | Day 274 to 280 |
| Week 41 | J | Day 281 to 287 |
| Week 42 | | Day 288 to 294 |
| Week 43 | | Day 295 to 301 |
| Week 44 | Day 306 to 312 | Day 302 to 308 |
| Week 45 | • | Day 309 to 315 |
| Week 46 | | Day 316 to 322 |
| Week 47 | | Day 323 to 329 |
| Week 48 | Day 334 to 340 | Day 330 to 336 |
| Week 49 | _ | Day 337 to 343 |
| Week 50 | | Day 344 to 350 |
| Week 51 | | Day 351 to 357 |
| Week 52 (EOSa) | Day 362 to 368* | Day 358 to 364 |
| Week 53 | • | Day 365 to 371 |
| Week 54 | | Day 372 to 378 |
| Week 55 | | Day 379 to 385 |
| Week 56 | Day 390 to 396 | Day 386 to 392 |
| Week 57 | | Day 393 to 399 |
| Week 58 | | Day 400 to 406 |
| Week 59 | | Day 407 to 413 |
| Week 60 | Day 418 to 424 | Day 414 to 420 |
| Week 61 | | Day 421 to 427 |
| Week 62 | | Day 428 to 434 |
| Week 63 | | Day 435 to 441 |
| Week 64 | Day 446 to 452 | Day 442 to 448 |
| Week 65 | | Day 449 to 455 |
| Week 66 | | Day 456 to 462 |
| Week 67 | | Day 463 to 469 |
| Week 68 | Day 474 to 480 | Day 470 to 476 |
| Week 69 | | Day 477 to 483 |
| Week 70 | | Day 484 to 490 |
| Week 71 | | Day 491 to 497 |
| Week 72 | Day 502 to 508 | Day 498 to 504 |
| Week 73 | | Day 505 to 511 |
| Week 74 | | Day 512 to 518 |
| Week 75 | - | Day 519 to 525 |
| Week 76 | Day 530 to 536* | Day 526 to 532 |
| Week 77 | | Day 533 to 539 |
| Week 78 | | Day 540 to 546 |
| Week 79 | | Day 547 to 553 |
| Week 80 | Day 558 to 564 | Day 554 to 560 |


| Week 81 | | Day 561 to 567 |
|-----------------|----------------|----------------|
| Week 82 | | Day 568 to 574 |
| Week 83 | | Day 575 to 581 |
| Week 84 | Day 586 to 592 | Day 582 to 588 |
| Week 85 | | Day 589 to 595 |
| Week 86 | | Day 596 to 602 |
| Week 87 | | Day 603 to 609 |
| Week 88 | Day 614 to 620 | Day 610 to 616 |
| Week 89 | | Day 617 to 623 |
| Week 90 | | Day 624 to 630 |
| Week 91 | | Day 631 to 637 |
| Week 92 | Day 642 to 648 | Day 638 to 644 |
| Week 93 | | Day 645 to 651 |
| Week 94 | | Day 652 to 658 |
| Week 95 | | Day 659 to 665 |
| Week 96 | Day 670 to 676 | Day 666 to 672 |
| Week 97 | | Day 673 to 679 |
| Week 98 | | Day 680 to 686 |
| Week 99 | | Day 687 to 693 |
| Week 100 | Day 698 to 704 | Day 694 to 700 |
| Week 101 | | Day 701 to 707 |
| Week 102 | | Day 708 to 714 |
| Week 103 | | Day 715 to 721 |
| Week 104 (EOSb) | Day 726 to 732 | Day 722 to 728 |

<sup>\*</sup>Note: At Weeks 24, 52 (EOSa), and 76, the WOMAC and Patient Global Assessment must be completed prior to the Week 24, 52 (EOSa), and 76 study medication injections, respectively.

# 17.2 Appendix 2 – Protocol Deviations Leading to Exclusion from Per-Protocol Analysis

| | Subjects Excluded from PPASB | | |
|---|---|---|---|
| Subject | Deviation | Category | Details |
| 0356016 | IP08 - Prohibited concomitant medication taken | Minor | SUBJECT RECEIVED 2 ML SYNVISC INJECTIONS IN TARGET KNEE 1X/WEEK FROM 25JUN2020 TO 09JUL2020 FOR OA KNEE PAIN. |
| | | Sub | jects Excluded from PPAS |
| Subject | Deviation | Category | Details |
| 0106017 | IP08 - Prohibited concomitant medication taken | Minor | OXYCODONE WAS TAKEN FROM 20NOV2019 TO 26NOV2019, 10 MG, PRN, ORAL ROUTE. |
| 0356001 | IP08 - Prohibited concomitant medication taken | Minor | SUBJECT TOOK HYDROCODONE-ACETAMINOPHEN, 5-325MG, PRN, FROM 04MAY-26MAY2019 AS TREATEMENT FOR AE OF KIDNEY STONES |
| 0356008 | DQ03 - Subject diary,<br>questionnaire, or patient<br>reported outcome<br>completion outside of<br>protocol requirements | Minor | SUBJECT WAS COMPLETING THE QUESTIONNAIRES ON THE INCORRECT TARGET KNEE FROM 21FEB2019 - 03JUL2019 DUE TO YPRIME PROGRAMMING ERROR. |
| 0356060 | IP08 - Prohibited concomitant medication taken | Minor | SUBJECT STARTED TAKING 20 MG OF AMITRIPTYLINE QD ORALLY ON 17OCT2019 FOR IRRITABLE BOWL SYNDROME AND CONMED IS ONGOING. |


| 4136003 | DQ03 - Subject diary,<br>questionnaire, or patient<br>reported outcome<br>completion outside of<br>protocol requirements | Minor | SUBJECT QUESTIONNAIRES WERE COMPLETED FOR THE INCORRECT TARGET KNEE FOR THE PERIOD OF 21FEB TO 11JU DUE TO YPRIME PROGRAMMING ERROR.(WEEK 4 - WEEK 24 VISITS WERE AFFECTED) |
|---|---|---|---|
| 1/1/36015 NCOL Subject non | | Major | SUBJECT HAD A KNEE ARTHROSCOPY IN TARGET KNEE (RIGHT) (PROHIBITED PER PROTOCOL), SUBJECT WAS ONLY HOSPITALIZED FOR 8 HOURS |
| 4266050 IP08 - Prohibited concomitant medication taken Major | | Major | CORTICOSTEROID INJECTION WAS ADMINISTERED INTRA-<br>ARTICULARLY INTO TARGET KNEE ON 23SEP2019. INJECTION<br>WAS RECEIVED ONCE WITH A DOSAGE OF 1ML |

<sup>\*\*</sup> Not excluded from PPAS entirely; however, efficacy data after this deviation will be censored, allowing for evaluation of both Phase A study injections with at least 12 weeks of follow-up.


# 17.3 Appendix 3 – Major Protocol Deviations and COVID-19 Protocol Deviations Not Associated with a Study Visit for Subjects in Phase B

| | | | | Date of<br>Week 52 | Counted as<br>Phase B |
|---|---|---|---|---|---|
| Subject | Deviation | Category | Details | Injection | <b>Deviation?</b> |
| | IP08 - Prohibited | | DUE TO COVID-19 AE, SUBJECT TOOK | | |
| 0356044 | concomitant | Minor | PREDNISONE 20 MG TABLET ORAL BID | 2020-05-22 | Yes |
| | medication taken | | FROM 28DEC2020 TO 01JAN2021 | | |
| 4136015 | NC01 - Subject<br>non-compliant<br>with protocol Major | | SUBJECT HAD A KNEE ARTHROSCOPY IN TARGET KNEE (RIGHT) (PROHIBITED PER PROTOCOL), SUBJECT WAS ONLY HOSPITALIZED FOR 8 HOURS [Dates from PROC: 22MAY2020] | 2020-07-09 | No |
| 4266050 IP08 - Prohibited concomitant medication taken Major | | Major | CORTICOSTEROID INJECTION WAS<br>ADMINISTERED INTRA-ARTICULARLY<br>INTO TARGET KNEE ON 23SEP2019.<br>INJECTION WAS RECEIVED ONCE WITH<br>A DOSAGE OF 1ML | 2020-05-26 | No |

# Signature Page for VV-TMF-183144 v0.0

| Reason for signing: Approved | Name: Jon Britt<br>Role: Manager, Biostatistics<br>Date of signature: 23-Sep-2021 04:45:48 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: Ismail Simsek<br>Role: Medical Director<br>Date of signature: 23-Sep-2021 14:37:51 GMT+0000 |
| Reason for signing: Approved | Name: Amy Halseth<br>Role: Executive Director, Clinical Science<br>Date of signature: 23-Sep-2021 15:17:57 GMT+0000 |
| Reason for signing: Approved | Name: Christopher Swearingen<br>Role: Vice President, Clinical Outcomes and<br>Analytics<br>Date of signature: 23-Sep-2021 15:27:13 GMT+0000 |

Signature Page for VV-TMF-183144 v0.0